CLINICAL TRIAL: NCT00341146
Title: Molecular Genetics Study of Nasopharyngeal Carcinoma: Characterization of NPC Susceptibility Gene(s)
Brief Title: Molecular Genetics Study of Nasopharyngeal Carcinoma: Characterization of NCP Susceptibility Gene(s)
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999902056; 02-C-N056
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2020-06-16 (Actual); Status verified 2020-06

CONDITIONS: Nasopharyngeal Carcinoma
Keywords: Cancer; Catonese Chinese; Genetic Predisposition; Genotyping; Triad analysis; Nasopharyngeal Cancer; NPC
MeSH Terms: conditions — Nasopharyngeal Carcinoma; Neoplasms; Genetic Predisposition to Disease; Nasopharyngeal Neoplasms

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Cross-Sectional

SUMMARY:
The objective of this study is to characterize genes associated either with susceptibility or resistance to the development nasopharyngeal carcinoma (NPC) in a Chinese population where the incidence of NPC is as high as 50 in 100,000. NPC has been and remains a unique model of human malignancy for understanding a multi-step carcinogenic process involving a ubiquitous virus (Epstein-Barr virus), environmental carcinogens, and an NPC susceptibility gene. Up to 95% of all NPC patients at early or late stage of the disease have IgA antibodies directed to the EBV virus VCA (viral capsid antigen). Environmental factors have also been implicated as significant risk factors in the development of NPC. In addition, certain alleles in HLA genes have shown associations with NPC, perhaps in concert with a family of T-cell receptor genes (TCR). Other data suggest that a microsatellite marker on Chromosome 6 may be associated with an NPC-disease associated gene.

DETAILED DESCRIPTION:
The objective of this study is to characterize genes associated either with susceptibility or resistance to the development nasopharyngeal carcinoma (NPC) in a Chinese population where the incidence of NPC is as high as 50 in 100,000. NPC has been and remains a unique model of human malignancy for understanding a multi-step carcinogenic process involving a ubiquitous virus (Epstein-Barr virus), environmental carcinogens, and an NPC susceptibility gene. Up to 95% of all NPC patients at early or late stage of the disease have IgA antibodies directed to the EBV virus VCA (viral capsid antigen). Environmental factors have also been implicated as significant risk factors in the development of NPC. In addition, certain alleles in HLA genes have shown associations with NPC, perhaps in concert with a family of T-cell receptor genes (TCR). Other data suggest that a microsatellite marker on Chromosome 6 may be associated with an NPC-disease associated gene.

We will use a "triad" approach to attempt to dissociate genetic from environmental and viral associations of NPC incidence. Blood samples will be collected from volunteers (probands) and family members (spouse and child and/or parent of patient) at two sites in Guangxi Province, China: the Cancer Research and Control Institute in Wuzhou City; and the Cang Wu County Cancer Hospital, located about 20 miles from Wuzhou. All cases will be EBV/IgA/VCA positive. These triad of samples will provide both control and haplotypic information on cases and controls. A database of pertinent clinical and family information will be created from a questionnaire filled in by hospital staff interviewers. Blood will be separated into plasma and peripheral blood mononuclear cells (PBMCs). Plasma will be tested at the Wuzhou Center for EBV/IgA/VCA. The PBMCs will be viably frozen and transported to the LGD at NCI/FCRDC, where they will be transformed into lymphoblastoid cell lines for extraction of DNA. At the LGD the DNAs will be screened for informative polymorphisms in candidate genes by DNA genotyping methods. Association analyses will be performed to detect linkages between informative polymorphisms in candidate genes by DNA genotyping methods. Association analyses will be performed to detect linkages between informative polymorphisms and clinical and family data. If a marker associated with development of NC is found, there are potential applications in diagnostics and therapy. Further, identification of allelic polymorphisms in genes with a role in NPC progression would offer definitive ties of such genes to the carcinogenic process.

Following this study, the samples will be maintained in our repository and curated through our central Laboratory database. Loss or destruction of these samples wil be recorded in our database and cannot impact the study participants in any way. We understand that studies subsequent to the completion of this protocol will require additional OHSR/IRB approval prior to commencement.

ELIGIBILITY:
* INCLUSION CRITERIA:

Individuals must meet the following eligibility criteria to be entered into the NPC study.

Cohort A: Proband: NPC positive (stage III or IV), age less than 50 at time of NPC diagnosis, and EBV/IgA/VCA positive. Spouse of Proband. Child of proband and of spouse (or a parent of the proband)

Cohort B: EBV/IgA/VCA positive 12 years ago and NPC negative. Spouse of proband. Child of proband and of spouse (or a parent of the proband).

EXCLUSION CRITERIA:

Persons with any of the following will be excluded from the study.

Persons who are unwilling or unable to given informed consent, or whose spouse and child(ren) (or parent) are willing to participate and give informed consent/assent.

Persons with no living spouse of child(ren)/parent.

Ages: 7 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Chinese population with a high incidence of NPC
Sampling Method: Non-Probability Sample
Enrollment: 6490 (Actual)
Dates: Start 2001-04-01 (Actual); Primary Completion 2006-08-20 (Actual); Study Completion 2006-09-20 (Actual)

PRIMARY OUTCOMES:
Collection from 9100 participants | 2006
  DNA Genotyping

CONTACTS AND LOCATIONS:
Overall Officials: Daniel W McVicar, Ph.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- Institute for Viral Disease Control & Prevention, Beijing, China

REFERENCES:
- [Background] O'Brien SJ, Nelson GW, Winkler CA, Smith MW. Polygenic and multifactorial disease gene association in man: Lessons from AIDS. Annu Rev Genet. 2000;34:563-591. doi: 10.1146/annurev.genet.34.1.563. PMID 11092839
- [Background] Zeng Y. Seroepidemiological studies on nasopharyngeal carcinoma in China. Adv Cancer Res. 1985;44:121-38. doi: 10.1016/s0065-230x(08)60027-5. No abstract available. PMID 2994402